CLINICAL TRIAL: NCT06176898
Title: The Effect of Neurostimulation on Patient Relevant Outcomes in Patients With Intermittent Claudication: a Pilot Study
Brief Title: Neurostimulation in Intermittent Claudication
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VS22/153016
Record Dates: First submitted 2023-09-26; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Claudication
Keywords: Vascular Medicine
MeSH Terms: conditions — Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neurostimulating device. (Experimental)
  Interventions: Device: Neurostimulating device

INTERVENTIONS:
Device: Neurostimulating device — A trained practitioner will apply the neurostimulator to the patient's ear. The patient will wear the neurostimulator for a period of three week with the position of the neurostimulator moving from one ear to the other on a weekly basis. After 3 weeks the neurostimulator will be removed and the patient will then undergo further clinical assessment at week 8.
  At the 8 week clinical assessment, the patient will undergo the same assessments, namely:
  * Six minute walking test (6MWT)
  * Quality of life assessment using both generic (Short form 12) and disease specific (Vascuqol) questionnaires

SUMMARY:
Intermittent claudication is a condition where a patient suffers with cramp-like pain experienced in the muscles of the legs (often the calf muscles) brought on by walking and relieved by stopping walking and resting. It is caused by furring of the arteries (atherosclerosis) often referred to as a circulation problem. It has a significant effect on a sufferers' quality of life. However, in 75% of patients with this condition, the leg symptoms will either stay static or improve slightly even with no treatment. The first line treatment is enrolment in an exercise / walking programme but these are not widely available on the NHS. Failing this, minimally invasive treatment - opening up the narrowing of the artery with either a balloon or stent - can be performed but they are not without risk (being an invasive treatment) and the narrowing often reoccurs in time. Due to the benign natural history of the leg, surgery is less frequently being used. This therefore leaves us with a large number of patients with symptoms with no treatment options and thus a poorer quality of life. Neurostimulation has been used to treat a number of neurological conditions. This study will use a specific device that is attached to the outer aspect of the ear to deliver a neurostimulation to a small branch of the Vagus nerve which through nerve pathways that course through the brain is believed to improve the blood supply to the lower legs.

DETAILED DESCRIPTION:
Lower limb peripheral arterial disease (PAD) is common, affecting over 200 million people worldwide and present in 12 to 14% of the global population (20% over the age of 75 years)1. The most common symptom is intermittent claudication, a symptom of muscular lower limb pain brought on by exertion and relieved by rest2.

PAD is the third leading cause of atherosclerotic cardiovascular morbidity, following coronary artery disease and stroke, yet the natural history of the limb in patients with IC is relatively benign with 75% of patients finding that symptoms either remain static or are somewhat improved with no treatment2. It is due to this natural history of the limb that there is an increasing tendency to manage patients with claudication conservatively (ie. Non-invasively).

In patients with intermittent claudication, CV prevention and exercise training are the cornerstones of management3. There is good evidence for enrolment of patients into a supervised exercise programme, providing bot improved walking distance and quality of life, yet widespread provision of such programmes are currently not available within the NHS and further are unlikely to be delivered within the coming years4.

Revascularisation has historically been indicated if daily life activity is severely compromised by the lower limb symptoms and such revascularisation is primarily performed endovascularly with balloon angioplasty +/- stent insertion where needed. The ability to perform endovascular revascularisation is determined by the anatomical location and severity of the lower limb atherosclerosis. Endovascular interventions work best with short focal stenoses rather than longer occlusion where surgical revascularisation is the better option2. Such interventions are invasive and carry risks including risk of amputation and so surgical revascularisation is now rarely performed for intermittent claudication. Further, there is now data available that suggests that early invasive revascularisation in patients with claudication may in the longer term increase the risk of major limb amputation. This means that there is a cohort of patients who have significant claudication symptoms affecting their quality of life who are either (i) not offered revasculairsation or (ii) not prepared to accept the risks of major lower limb revascularisation.

Given this, there is a need to explore further non-invasive methods that could enhance walking distances in patients with IC and thus improve overall quality of life and overall cardiovascular fitness without exposing patients to invasive revascularisations.

There has been an increasing focus on the role of neuromodulation in the management of several chronic diseases5. Neuromodulation is defined as a physiological process which consists of the alteration of neuronal and synaptic properties by neurons or substances released by neurons. Neuromodulation, thanks to intrinsic and extrinsic brain feedback loops, seems to be the best way to exploit brain plasticity for therapeutic purposes.

Vasomotion is believed to play a pivotal role in capillary function and microcirculation. Based on spontaneous oscillating change of arteriole and venule diameter it has been theoretically suggested that oscillatory perfusion may be superior to steady-state flow. It has been shown that continuous electrical stimulation of sympathetic nerves induces a tonic vasoconstriction6.

Consistently, procedures like lumbar sympathectomy are used to enhance blood supply in malperfused limbs. Enhanced parasympathetic stimulation may also cause vasodilatation. We hypothesise that auricular vagus stimulation could modulates afferent parasympathetic activity and potentially improves microcirculation7.

From a medical viewpoint, neurostimulation techniques do provide several advantages with respect to conventional drug or invasive surgical treatments:

* Specificity: stimulation can be targeted to particular areas avoiding the insurgence of systemic side-effects, typical of traditional drug therapies;
* Safety: neurostimulation techniques are generally well-tolerated and almost devoid of dangerous side effects;
* Flexibility: the treatment can be interrupted at any time. One such device that allows neurostimulation to be delivered is the DUCEST neurostimulator device. This is a minimally invasive device that stimulates the afferent branches of the vagus nerve situated within the outer aspect of the ear lobe. (Fossa triangularis).

Figure 1: Anatomical landmarks within the ear.

Figure 2: The Ducest Medical device.

Figure 3: The application of the Ducest Medical device to the ear.

One study in the UK has looked at the effect of the DUCEST neurostimulator in 30 patients with the most severe limb ischaemia who had no revascularisation option and has found that were significant improvements in the size of and flow through the calf arteries. This corresponded with an avoidance in major limb amputation in 11 of the 30 patients.

No study in the UK has formally assessed the effect of such an intervention on patients with IC.

There is a large cohort of patient who would potentially benefit from a low risk, non-invasive intervention aimed at increasing walking distances and improving quality of life.

ELIGIBILITY:
Inclusion Criteria:

* • Rutherford b/c intermittent claudication with stable symptoms for 6 months with a decision not to undergo any revascularization.

Exclusion Criteria:

* • Critical limb ischaemia

  * Previous external ear surgery
  * Patients with either a cochlear implant or a permanent pacemaker / cardiac defibrillator device
  * Significant cardiorespiratory or musculoskeletal disease (as determined by the medical team) that would contraindicate a 6-minute walk test

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal walking distance determined from the six-minute walk test | At baseline and at 8 weeks
  Maximal walking distance determined from the six-minute walk test (6MWT)

SECONDARY OUTCOMES:
Quality of life analysis using both generic and disease specific quality of life | At baseline and at 8 weeks
  Quality of life analysis using both generic and disease specific quality of life, using quality of life questionnaire
Patient acceptance of the neurostimulator device | At baseline and at 8 weeks
  Patient acceptance of the neurostimulator device using questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No